CLINICAL TRIAL: NCT01189864
Title: Collagen Crosslinking With Ultraviolet-A in Asymmetric Corneas
Brief Title: Cross-linking of Corneal Collagen (CXL) With Ultraviolet-A in Asymmetric Corneas
Status: Terminated | Type: Observational
Why Stopped: Terminated to initiate FDA IND-cleared study protocol
Sponsor: Cxlusa (Industry)
Responsible Party: Sponsor
Other Study IDs: CXL (12 & older)
Record Dates: First submitted 2010-07-20; First posted 2010-08-27 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Keratoconus; Ectasia; Degeneration
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic | interventions — Moxifloxacin; Ketorolac Tromethamine; Ketorolac; Steroids; Fluorometholone; prednisolone acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Ciprofloxicin or Vigamox or other.
  Interventions: Drug: Ciprofloxicin or Vigamox or other.
- Nonsteroidal (Acular, Voltaren Xibrom, etc)
  Interventions: Drug: Nonsteroidal (Acular, Acuvail, Voltaren Xibrom, etc)
- Steroid (FML, Pred Forte, Flarex, etc.)
  Interventions: Drug: Steroid (FML, Pred Forte, Flarex, etc.)

INTERVENTIONS:
Drug: Ciprofloxicin or Vigamox or other. — Ciprofloxicin or Vigamox or other to be used qid till epithelialized.
  Groups: Ciprofloxicin or Vigamox or other.
Drug: Nonsteroidal (Acular, Acuvail, Voltaren Xibrom, etc) — Nonsteroidal (Acular, Voltaren Xibrom, etc) qid up to 5-10 days post-op
  Groups: Nonsteroidal (Acular, Voltaren Xibrom, etc)
Drug: Steroid (FML, Pred Forte, Flarex, etc.) — Steroid (FML, Pred Forte, Flarex, etc.) to be used qid to qd for 1-8 weeks.
  Groups: Steroid (FML, Pred Forte, Flarex, etc.)

SUMMARY:
The purpose of this study is to evaluate the efficacy of ultraviolet-A (UVA)-induced cross-linking of corneal collagen (CXL) as a method to increase the biomechanical and biochemical stability of the cornea by inducing additional cross-links within or between collagen fibers using UVA light and the photo- mediator riboflavin. The purpose of this study is to generate data for presentation at medical meetings and for peer-review publication. The data generated by this study will not be submitted to the FDA to support commercialization of these riboflavin drops.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older
* Diagnosis of keratoconus, FFKC, post-LASIK ectasia, or pellucid marginal degeneration or forme fruste pellucid marginal degeneration (FFPMD).
* Diagnosis of FFKC
* History of Radial Keratotomy with fluctuating vision
* Ability to provide written informed consent
* Likely to complete all study visits
* Minimum corneal thickness of at least 300 Measured by ultrasound or Pentacam
* At least 6 months since last corneal surgery (Intacs/PRK/LASIK/Epi-LASIK/LASEK)

Exclusion Criteria:

* Severe corneal scarring that markedly affects vision
* Contraindications to any study medications or their components
* Pregnancy or breast feeding
* Active Herpes Corneal Disease

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic.
Sampling Method: Probability Sample
Enrollment: 3493 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2017-02-03 (Actual); Study Completion 2017-02-03 (Actual)

PRIMARY OUTCOMES:
Increase the biomechanical and biochemical stability of the cornea by inducing additional cross-links within | 1 year

SECONDARY OUTCOMES:
increase the biomechanical and biochemical stability of the cornea between collagen fibers using UVA light and the photo- mediator riboflavin | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: William Trattler, MD, Principal Investigator — The Center for Excellence in Eye Care; Jodi Luchs, MD, Principal Investigator — South Shore Eye Care LLP; Shamik Bafna, MD, Principal Investigator — Cleveland Eye Clinic; Parag Majmudar, MD, Principal Investigator — Chicago Cornea Consultants, LTD; Jay Schwartz, MD, Principal Investigator — Schwartz Laser Eye Center; Jonathan Davidorf, MD, Principal Investigator — Davidorf Eye Group; Daniel Goodman, MD, Principal Investigator — Goodman Eye Center; Jonathan Talamo, MD, Principal Investigator — Talamo Laser Eye Center; Sandy Feldman, MD, Principal Investigator — Clear View Eye & Laser Medical Center; Gregg Berdy, MD, Principal Investigator — Ophthalomology Associates; Lance Forstot, Principal Investigator — Corneal Consultants of Colorado, P.C; Mark Kontos, MD, Principal Investigator — Empire Eye Physicians; Audrey Rostov, MD, Principal Investigator — Northwest Eye Surgeons; John Hovanesian, MD, Principal Investigator — Harvard Eye Associates
Locations (16):
- United States (16):
  - Schwartz Laser Eye Center, Scottsdale, Arizona
  - Harvard Eye Associates, Laguna Hills, California
  - Clear View Eye & Laser Medical Center, San Diego, California
  - San Francisco, California
  - Davidorf Eye Group, West Hills, California
  - Corneal Consultants of Colorado, P.C, Littleton, Colorado
  - The Center for Excellence in Eye Care, Miami, Florida
  - Chicago Cornea Consultants, LTD, Hoffman Estates, Illinois
  - TLC Laser Eye Center, Rockville, Maryland
  - Talamo Laser Eye Center, Waltham, Massachusetts
  - Ophthalomology Associates, St Louis, Missouri
  - South Shore Eye Care LLP, Wantagh, New York
  - Cleveland Eye Clinic, Brecksville, Ohio
  - TLC Laser Eye Center, Fairfax, Virginia
  - Northwest Eye Surgeons, Seattle, Washington
  - Empire Eye Physicians, Spokane Valley, Washington